CLINICAL TRIAL: NCT04041531
Title: Determination of the Oxygen Dissociation Curve Under the Conditions of an Avalanche Burial With an Air Pocket
Brief Title: Triple H ODC Trial
Acronym: 3H-ODC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 1123/2019
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hypoxia; Hypothermia, Accidental; Hypercapnia; Avalanche, Landslide, or Mudslide
MeSH Terms: conditions — Hypoxia; Hypothermia; Hypercapnia | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 16 combinations of 4 levels of pCO2 and 4 levels of temperature will be assessed for each participant
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — venous blood sampling for oxygen affinity in-vitro test

SUMMARY:
In an avalanche burial with an air pocket hypercapnia (and hypoxia) develops within few minutes, hypercapnia increases the rate of cooling and therefore the development of hypothermia. The Triple H Syndrome (Hypoxia, Hypercapnia, Hypothermia) occurs. This specific combination of the three parameters is unique for avalanche burial with an air pocket. Every single parameter has a substantial effect on the hemoglobin-oxygen dissociation curve, but until now no study described the combination of these three parameters. This curve will be measured under these specific conditions in a specifically developed in vitro model, to quantify its shifts and to show if there are combined effects of pCO2 and temperature. The newly developed method will be validated in comparison with an established method. The project will be performed with whole blood, drawn by healthy volunteers, in an experimental setting. The samples will be blinded to the investigator and analyzed in a randomized manner.

DETAILED DESCRIPTION:
The ODC is a function of pO2 and SO2. pO2, the independent variable, is plotted on the x axis, SO2 on the y axis. For the determination of this function, a pairwise measurement of pO2 and the corresponding SO2 is to be performed. Using nonlinear regression analysis, the ODC can be fitted to the measured points that describe the relation of pO2 and SO2 and characteristic parameters like p50 value and inflection points can be calculated.

To measure the ODC under the conditions of the Triple H Syndrome (Hypoxie, Hypercapnia, Hypothermia), the temperature and the pCO2 have to be changed and controlled during the measurement. No commercially available instrument is able to obtain this. Therefore, we envisaged the development of an entirely new approach.

In the 3H ODC trial venous blood will be drawn from 18 - 40 years old female and male volunteers by a unique venipuncture. The participants have to be in a fasted situation, ASA I and nonsmokers. The blood sample will be immediately pseudonymized and stored on ice and a venous blood gas analysis will be carried out (pH, Hb, COHb, MetHb, FHb). Simultaneous to the main measurement, 2,3 BPG will be quantified by an ELISA test and any unknown hemoglobinopathy will be excluded by Hemoglobin Electrophoresis. In the 3H ODC trial 4 different pCO2 levels and 4 different temperatures will be analyzed in the resulting 16 combinations. In each round a lot of ODCs will be measured, the measurement chamber will be filled with participants blood samples in a randomized manner. After the measurements, the blood samples will be discarded.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* fasted situation
* ASA I
* Informed Consent

Exclusion Criteria:

* any drug abuse
* any drug intake within the last 10 days
* smoking
* known hemoglobinopathy
* relevant illness within last 14 days
* relevant blood loss within last 14 days
* pregnancy or breast-feeding
* participation in any pharmacological study
* exposure to high altitude (> 3000 m) within last 4 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
amount of p50 in different levels of hypercapnia and hypothermia | day 1
  amount of p50 in mmHg (p50 = pO2 when oxygen saturation of hemoglobin is 50%)

SECONDARY OUTCOMES:
amount of p50 shift due to sex | day 1
  amount of p50 in mmHg (p50 = pO2 when oxygen saturation of hemoglobin is 50%)
amount of inflection point in different levels of hypercapnia and hypothermia | day 1
  amount of inflection point in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ströhle, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- General and Surgical Critical Care Medicine, Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No